CLINICAL TRIAL: NCT04852120
Title: A Post-marketing Drug Intensive Monitoring Study of Compound Sodium Picosulfate Granules for Bowel Preparation in Chinese Population
Brief Title: Compound Sodium Picosulfate Granules for Bowel Preparation in Chinese Population
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: DeltaMed (Industry)
Responsible Party: Sponsor
Other Study IDs: 000373
Record Dates: First submitted 2021-03-25; First posted 2021-04-21 (Actual); Results first posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-07

CONDITIONS: Bowel Cleansing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Compound Sodium Picosulfate Granules
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Compound Sodium Picosulfate Granules administered by the patient prior to X-ray examination, endoscopy or surgery when judged clinically necessary in accordance to usual practice consistent with the local prescribing information.

SUMMARY:
High-quality bowel preparation plays an important role in ensuring a safe and successful X-ray examination, endoscopy or some kinds of bowel surgeries. Inadequate bowel preparation may lead to incomplete examination of the colonic mucosa, may require increased operation time and difficulty, and incur the costs for rescheduling or performing other examinations. Early attention to the influencing factors of bowel cleansing effect and taking positive measures can effectively improve the success rate and diagnosis rate of endoscopic and radiological examinations, and reduce the possibility of postoperative complications and local infections. In 2019, China released the latest "Guidelines for Bowel Preparation Related to Digestive Endoscopy", emphasizing the importance of dietary restrictions and patient notification and education. The "Guideline" also recommends that sodium picosulfate, magnesium oxide, and anhydrous citric acid can be used for bowel preparation before endoscopy and is well tolerated (recommended strength: weak; evidence quality: moderate). The other used colonic cleansing agents also include polyethylene glycol (PEG) electrolyte powder, magnesium salt, sodium phosphate, mannitol and Chinese herbal medicine. Each carries its own properties, indications and safety profiles.

Compound Sodium Picosulfate Granules is a compounded preparation consisting of sodium picosulfate and magnesium citrate. Each sachet contains 10 mg of sodium picosulfate, 3.5 g of magnesium oxide and 12.0 g of citric acid. It is white to slightly yellow crystalline powder, with a slight orange flavour. Sodium picosulfate is transformed by colonic bacteria to form an active metabolite: bis-(p-hydroxyphenyl)-pyridyl-2-methane, Bis-(p-hydroxyphenyl)-pyridyl-2-methane (BHPM), which acts directly on the colonic mucosa to stimulate colonic peristalsis. Magnesium oxide and citric acid react to create magnesium citrate (when dispersed in a solution), which is an osmotic agent that causes water to be retained within the gastrointestinal tract. The stimulant laxative activity of sodium picosulfate together with the osmotic laxative activity of magnesium citrate produces a purgative effect, which can be used to clean the bowel prior to X-ray examination, endoscopy or bowel surgery.

Since its first marketing in the United Kingdom (UK) in December 1980, Compound Sodium Picosulfate Granules has been approved in more than 80 countries and regions, including Germany (2010), France (2010), Spain (2011), Italy (2011), United States (2012) and Japan (2016), under the tradename PICOLAX, PICOPREP or PREPOPIK. In 2018, Compound Sodium Picosulfate Granules was officially approved in China with the indication: for preparation of bowel cleansing prior to X-ray examination, endoscopy or surgery when judged clinically necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been prescribed Ferring Compound Sodium Picosulfate Granules
* Agree to participate in this study and sign the informed consent form (ICF).

Exclusion Criteria:

- Patients who are enrolled in other on-going studies, which prohibit any participation in this non-interventional study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been prescribed Ferring Compound Sodium Picosulfate Granules at the participating sites will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (8):
- China (8):
  - Ferring Investigational Site, Beijing
  - Ferring Investigational Site, Dalian
  - Ferring Investigational Site, Fuzhou
  - Ferring Investigational Site, Jingdezhen
  - Ferring Investigational Site, Nanjing
  - Ferring Investigational Site, Ningbo
  - Ferring Investigational Site, Qiqihar
  - Ferring Investigational Site, Xi'an

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed in 14 investigational sites in China between April 2021 and December 2022
Pre-assignment Details: In total, 3000 participants were screened and enrolled.
Period: Overall Study
Arm/Group | Compound Sodium Picosulfate Granules
Started | 3000
Completed | 3000
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Compound Sodium Picosulfate Granules
Number analyzed (Participants) | 3000
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 2700
  >=65 years | 292
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.99 (13.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1546
  Male | 1454
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3000
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 3000
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.16 (3.22)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Known Adverse Drug Reactions (ADRs)
Description: An adverse drug reaction (ADR) is characterized by the suspicion of a causal relationship between the medicine and the occurrence, i.e. judged as being at least possibly related to treatment by the reporter or a reviewing health professional.
  An ADR is a response to a medicinal product which is noxious and unintended. This includes adverse reactions which arise from:
  * The use of a medical product within the terms of the marketing authorization;
  * The use outside the terms of the marketing authorization, including overdose, off-label use, misuse, abuse and medication errors;
  * Occupational exposure.
Time Frame: Up to 37(+2) hours after drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Compound Sodium Picosulfate Granules
Number analyzed (Participants) | 3000
Participants
  Abdominal Pain | 2
  Dizziness | 1
  Nausea | 2
  Vomiting | 6

2. Primary Outcome: Occurrence of Unexpected Adverse Events (AEs)/ADRs
Description: Adverse event (AE) is any untoward medical condition or the deterioration of a pre-existing medical condition in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
  Unexpected adverse reaction refers to a drug reaction whose nature, severity, specificity, or outcome is not consistent with the term or description listed in the current local/regional label. This includes events that may be symptomatically and pathophysiological related to an event listed in the labelling but differ from the event because of greater severity or specificity.
Time Frame: Up to 37(+2) hours after drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Compound Sodium Picosulfate Granules
Number analyzed (Participants) | 3000
Participants
  Abdominal Distension | 1
  Abnormal Faeces | 1
  Amaurosis | 1
  Asthenia | 1
  Chest Discomfort | 1
  Dizziness | 1
  Palpitations | 1
  Syncope | 1

3. Primary Outcome: Incidence and Risk Factors of Serious Adverse Events (SAEs)/Serious Adverse Drug Reactions (SADRs)
Description: The incidence below is Syncope.
  A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose that:
  * Results in death
  * Is life-threatening
  * Is a congenital anomaly/birth defect
  * Results in persistent or significant disability/incapacity
  * Results in unplanned inpatient hospitalisation or prolongation of existing hospitalisation
  * Is an important medical event that may jeopardise the participant or may require intervention to prevent one of the outcomes listed above
Time Frame: Up to 37(+2) hours after drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Compound Sodium Picosulfate Granules
Number analyzed (Participants) | 3000
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from signing the informed consent form (ICF) to about 37(+2) hours after first medication.
Arm/Group | Compound Sodium Picosulfate Granules
All-Cause Mortality (participants affected / at risk) | 0/3000
Serious Adverse Events (participants affected / at risk) | 1/3000
Other Adverse Events (participants affected / at risk) | 0/3000
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Compound Sodium Picosulfate Granules (N=3000)
Syncope (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT04852120/Prot_SAP_000.pdf